CLINICAL TRIAL: NCT01503814
Title: Simplified Cardiovascular Management Study: A Cluster-Randomized Trial to Evaluate the Effects of a Simplified Cardiovascular Management Program in Tibet, China and Haryana, India
Brief Title: Simplified Cardiovascular Management Study
Acronym: SimCard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03COE-RA02; HHSN268200900027C (Other Grant/Funding Number: NHLBI)
Record Dates: First submitted 2011-12-30; First posted 2012-01-04 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2014-08

CONDITIONS: Cardiovascular Disease
Keywords: hypertension; primary care; cardiovascular disease prevention; high cardiovascular risk; diuretics; aspirin; smoking cessation; salt reduction; Tibet
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Usual Care) (No Intervention): Control
- Intervention (Experimental): Use of a simplified guideline-based CVD prevention and management scheme by village doctors targeting high risk individuals focusing on a"2+2"model: 2 therapeutic lifestyle recommendations (smoking cessation and salt consumption reduction) plus prescription of 2 low-cost drugs (aspirin and low-dose diuretics) when applicable
  Interventions: Other: Simplified cardiovascular disease management

INTERVENTIONS:
Other: Simplified cardiovascular disease management — This study is a complex pragmatic trial.The intervention includes a "package" of 4 main established measures for cardiovascular prevention and management:
  2 therapeutic lifestyle recommendations- smoking cessation (if applicable) and reduced salt consumption
  2 drug therapies (if applicable)- hydrochlorothiazide, 25mg tab, 1/2 tab daily (12.5mg/day) and aspirin, 25mg tab, 3 tabs daily (75mg/day)
  Arms: Intervention

SUMMARY:
The goal of this study is to develop, pilot test, and evaluate a highly simplified but guideline-based program for cardiovascular management for application in resource-scarce settings. The study aims to assess the effects of implementing a simple low-cost cardiovascular management program for high-risk individuals, delivered by primary care providers (PCPs) or community health workers (CHWs), on the proportion of patients appropriately treated with diuretics as well as a number of secondary outcomes in resource-scarce Tibet, China and Haryana India.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of morbidity, mortality, and disability in not only developed, but also developing countries. There are well-established interventions such as lifestyle modification and drug therapies, i.e., aspirin and low-dose diuretics, that along with their consistent use, can help alleviate these burdens if the practicalities of how to deliver such care to large numbers in resource-poor settings at low cost can be resolved. One particular cost-effective approach for secondary prevention of CVD is to identify and manage individuals at high CVD risk in order to prevent or delay events. This approach has been tested in the rural Andhra Pradesh Cardiovascular Prevention Study in India and is currently being implemented in rural areas of northern China in the China Rural Health Initiative funded by NHLBI.

This project aims to address the highly prevalent problem of CVD in even more remote and poor areas of China and India that have received only minimal attention so far, specifically Tibet, China and Haryana, India. This pilot project will be a cluster-randomized controlled interventional trial that will include a total of 15 villages in 6 townships in Gongbujiangda County and 12 villages in 6 townships in Linzhou County in Tibet, China and 12 villages in the state of Haryana in India. The study will last for one year. The villages will be randomized to receive either the intervention package or usual care. At baseline, village-wide screenings will be done to identify high-risk individuals in the selected villages who will then be followed throughout the study to about one year.

The interventional model will make use of a highly simplified cardiovascular disease management plan targeting lifestyle modification and utilization of basic drug regimens to help overcome the barriers in prevention and management of CVD in these areas with extremely limited economic and natural resources, minimal public awareness to the problem, and a lack of trained healthcare professionals.

Electronic blood pressure monitors will be used in all villages to measure the blood pressures of these individuals. However accuracy of the electronic blood pressure monitor measurements needs to be considered due to Tibet's high altitude. A study to validate and calibrate the selected blood pressure monitor model in both plains and high altitude areas will thus be undertaken using the validation procedure published by the European Society of Hypertension (ESH) to ensure accuracy.

ELIGIBILITY:
Inclusion Criteria:

Age is equal or older than 40 years old AND the subject has a self-reported history of ANY of the following diseases:

* CVD OR
* Diabetes OR
* Stroke (including both Ischemic Stroke and Haemorrhagic Stroke) OR
* Measured systolic blood pressure is equal or greater than 160mmHg at two different time points in the same day during the baseline survey.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2086 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Net Difference in Proportion Treated with Low-dose Diuretics | baseline and at one year
  The primary outcome will be the net differences between the changes in the proportion of high-risk individuals treated with low-dose diuretics pre-and-post intervention between intervention and control villages. The outcome measure will be assessed via a questionnaire that will ask about low-dose diuretics usage that will be administered at baseline and then again following the intervention period at around one year.

SECONDARY OUTCOMES:
Net Difference from Baseline in Mean Blood Pressure | baseline and at one year
  The net difference in mean post-intervention blood pressure changes of high-risk patients from baseline between intervention and control villages will be measured. This outcome measure will be taken at baseline and then again following the intervention period at around one year using a standardized electronic blood pressure monitor. Each subject's blood pressure will be taken twice at different time points within the same visit for the baseline measurement and one year follow-up measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Lijing Yan, PhD, Principal Investigator — The George Institute, China (Beijing, CN)
Locations (3):
- China (2):
  - Linzhou, Lhasa, Tibet
  - Gongbujiangda, Linzhi, Tibet
- Faridabad, Haryāna, India

REFERENCES:
- [Background] Oakley A, Strange V, Bonell C, Allen E, Stephenson J; RIPPLE Study Team. Process evaluation in randomised controlled trials of complex interventions. BMJ. 2006 Feb 18;332(7538):413-6. doi: 10.1136/bmj.332.7538.413. PMID 16484270
- [Background] Manuel DG, Lim J, Tanuseputro P, Anderson GM, Alter DA, Laupacis A, Mustard CA. Revisiting Rose: strategies for reducing coronary heart disease. BMJ. 2006 Mar 18;332(7542):659-62. doi: 10.1136/bmj.332.7542.659. PMID 16543339
- [Background] O'Brien E, Pickering T, Asmar R, Myers M, Parati G, Staessen J, Mengden T, Imai Y, Waeber B, Palatini P, Gerin W; Working Group on Blood Pressure Monitoring of the European Society of Hypertension. Working Group on Blood Pressure Monitoring of the European Society of Hypertension International Protocol for validation of blood pressure measuring devices in adults. Blood Press Monit. 2002 Feb;7(1):3-17. doi: 10.1097/00126097-200202000-00002. No abstract available. PMID 12040236
- [Background] World Health Organization. Global strategy on diet, physical activity and health, F.-S.W.H. Assembly, Editor. 2004: Available from: http://www.who.int/dietphysicalactivity/goals/en/index.html.
- [Background] Murray C, and Lopez A. The Global Burden of Disease: A Comprehensive Assessment of Mortality and Disability from Disease, Injuries and Risk Factors in 1990 and Projected to 2020. Boston, Mass: Harvard School of Public Health., 1996.
- [Background] Yusuf S, Reddy S, Ounpuu S, Anand S. Global burden of cardiovascular diseases: part I: general considerations, the epidemiologic transition, risk factors, and impact of urbanization. Circulation. 2001 Nov 27;104(22):2746-53. doi: 10.1161/hc4601.099487. PMID 11723030
- [Background] China guideline of hypertension updated 2005 Progression in the diagnosis and management of hypertension. China Hypertension League, 2005.
- [Background] Li SS, Zhao XS, Ba S, He F, Ke L, Li N, Yan LL, Wu YF. (2009, November). Validation of electronic sphygmomanometers against mercury sphygmomanometers at high altitude in Tibet. Poster presented at The Word Hypertension Congress 2009.
- [Background] National Vascular Disease Prevention Alliance, Guidelines for the Assessment of Absolute Cardiovascular Disease Risk. 2009, National Heart Foundation of Australia: Melbourne.
- [Derived] Tian M, Yin X, Dunzhu D, Liu Z, Li C, Sun H, Song C, Sangzhu L, Patel A, Redfern J, Yan LL. A qualitative evaluation of a simplified cardiovascular management program in Tibet, China. Global Health. 2018 Mar 1;14(1):24. doi: 10.1186/s12992-018-0342-0. PMID 29490675
- [Derived] Tian M, Ajay VS, Dunzhu D, Hameed SS, Li X, Liu Z, Li C, Chen H, Cho K, Li R, Zhao X, Jindal D, Rawal I, Ali MK, Peterson ED, Ji J, Amarchand R, Krishnan A, Tandon N, Xu LQ, Wu Y, Prabhakaran D, Yan LL. A Cluster-Randomized, Controlled Trial of a Simplified Multifaceted Management Program for Individuals at High Cardiovascular Risk (SimCard Trial) in Rural Tibet, China, and Haryana, India. Circulation. 2015 Sep 1;132(9):815-24. doi: 10.1161/CIRCULATIONAHA.115.015373. Epub 2015 Jul 17. PMID 26187183
- [Derived] Ajay VS, Tian M, Chen H, Wu Y, Li X, Dunzhu D, Ali MK, Tandon N, Krishnan A, Prabhakaran D, Yan LL. A cluster-randomized controlled trial to evaluate the effects of a simplified cardiovascular management program in Tibet, China and Haryana, India: study design and rationale. BMC Public Health. 2014 Sep 6;14:924. doi: 10.1186/1471-2458-14-924. PMID 25194850